CLINICAL TRIAL: NCT02565953
Title: Primary Patency in Post-angioplasty Dysfunctional Arteriovenous Fistula in Renal Dialysis: Paclitaxel-releasing PTA Balloon Catheter vs PTA Balloon
Acronym: FISBAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FISBAL
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2017-03

CONDITIONS: Arteriovenous Fistula Renal Dialysis Devices Obstruction
Keywords: Vascular access devices obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel-releasing PTA balloon catheter (Experimental): Treatment of renal dialysis arteriovenous fistula stenosis with paclitaxel-releasing percutaneous transluminal angioplastic (PTA) balloon catheter.
  Interventions: Device: Paclitaxel-releasing PTA balloon catheter
- PTA Balloon catheter (Active Comparator): Treatment of renal dialysis arteriovenous fistula stenosis with percutaneous transluminal angioplastic (PTA) balloon catheter.
  Interventions: Device: PTA balloon catheter

INTERVENTIONS:
Device: Paclitaxel-releasing PTA balloon catheter
  Arms: Paclitaxel-releasing PTA balloon catheter
Device: PTA balloon catheter
  Arms: PTA Balloon catheter

SUMMARY:
In recent years the use of paclitaxel releasing percutaneous transluminal angioplastic (PTA) balloon catheter is spreading in vascular pathology, mainly in stenosis infrainguinal arteries. This device combined the mechanical action of PTA balloon with the antiproliferative effects of paclitaxel. The use of these devices in venous pathology is limited. This devices could improve the treatment of renal dialysis arteriovenous fistula stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal dialysis with arteriovenous fistula (AVF) at least 3 months before.
* Patient diagnosed with AVF stenosis by clinical and radiological criteria
* Sign informed consent

Exclusion Criteria:

* Pregnant or breastfeeding
* Patients with AVF stenosis not could be treated with PTA catheter
* Paclitaxel allergy
* Iodinated contrast allergy
* Local or systemic active infection
* Life expectancy less than 12 moths

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Freedom from target lesion revascularization | 12 months
  Percentage of patients that do not need any revascularization proceeding during the following twelve months after catheter insertion.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario Puerto Real, Puerto Real, Cádiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Juan Ramón Jiménez, Huelva